CLINICAL TRIAL: NCT07341867
Title: A Pilot Study of Duffy Null-Specific Dose Modifications for Individuals With Duffy Null Phenotype Receiving Standard of Care Systemic Anti-Cancer Therapies
Brief Title: Systemic Anti-Cancer Therapy Dose Modifications for Individuals With Duffy Null Phenotype
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew Hantel, MD (Other)
Responsible Party: Sponsor-Investigator, Andrew Hantel, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-555
Record Dates: First submitted 2025-12-15; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma; Triple Negative Breast Cancer; Duffy Blood Group, Chemokine Receptor Gene Mutation; Duffy Blood Group, Chemokine Receptor Gene C.-67T>C
Keywords: Duffy Null Phenotype; Multiple Myeloma; Triple Negative Breast Cancer; Dosing guidelines
MeSH Terms: conditions — Multiple Myeloma; Triple Negative Breast Neoplasms | interventions — Dexamethasone; Calcium Dobesilate; Bortezomib; Lenalidomide; daratumumab; Carboplatin; Paclitaxel; pembrolizumab; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Multiple myeloma (MM) (Experimental): Participants with Multiple Myeloma and identified Duffy Null phenotype will receive standard of care (Dara-RVD) per institutional protocol with dosage adjustments per Duffy-Null guidance.
  Study treatment cycle lasts 28 days
  * dexamethasone 1X daily on days 1, 2, 8, 9, 15, 16, 22, 23 for 6 cycles
  * lenalidomide 1x daily on days 1-21 for 6 cycles
  * bortezomib 1x weekly for 2 cycles
  * daratumumab 1x weekly up to 2 cycles, then every 14 days for 4 more cycles
  Interventions: Drug: Dexamethasone; Drug: Bortezomib; Drug: LENALIDOMIDE; Drug: Daratumumab
- Arm B: Triple-Neg Breast Cancer (Experimental): Participants with Triple Negative Breast Cancer and identified Duffy Null phenotype will receive standard of care (Keynote-522) per institutional protocol with dosage adjustments per Duffy-Null guidance
  Study treatment cycle lasts 21 days
  * Pembrolizumab 1x every 21 days on day 1 for cycles 1-4
  * Paclitaxel 1x weekly on D1, 8, and 15 for cycles 1-4
  * Carboplatin 1x weekly on D1, 8, and 15 for cycles 1-4
  * Doxorubicin 1x every 14 days for cycles 5-8
  * Cyclophosphamide 1x every 14 days for cycles 5-8
  * Pembrolizumab 1x every 21 days on day 1 for cycles 5-8
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Pembrolizumab; Drug: Cyclophosphamide; Drug: Doxorubicin

INTERVENTIONS:
Drug: Dexamethasone — Tablet, taken orally
  Other Names: Decadron; Dexamethasone Intensol; Dexasone; Solurex; Baycadron
  Arms: Arm A: Multiple myeloma (MM)
Drug: Bortezomib — Intravenous infusion
  Other Names: Velcade
  Arms: Arm A: Multiple myeloma (MM)
Drug: LENALIDOMIDE — Tablet, taken orally
  Other Names: Revlimid
  Arms: Arm A: Multiple myeloma (MM)
Drug: Daratumumab — Intravenous infusion
  Other Names: Darzalex; Darzalex Faspro
  Arms: Arm A: Multiple myeloma (MM)
Drug: Carboplatin — Intravenous infusion
  Other Names: Paraplatin
  Arms: Arm B: Triple-Neg Breast Cancer
Drug: Paclitaxel — Intravenous infusion
  Other Names: Taxol
  Arms: Arm B: Triple-Neg Breast Cancer
Drug: Pembrolizumab — Intravenous infusion
  Other Names: Keytruda; Keytruda Qlex
  Arms: Arm B: Triple-Neg Breast Cancer
Drug: Cyclophosphamide — Intravenous infusion
  Other Names: Cytoxan
  Arms: Arm B: Triple-Neg Breast Cancer
Drug: Doxorubicin — Intravenous infusion
  Other Names: Adriamycin; Rubex; Doxorubicin hydrochloride (HCl); Hydroxydaunorubicin; ADM
  Arms: Arm B: Triple-Neg Breast Cancer

SUMMARY:
This study is comprised of a main study, an observational study, and optional survey studies. The main study is being done to see whether using Duffy null specific treatment dosing guidelines can reduce or delay dose modifications and avoid neutropenic fever (fever in the setting of low neutrophils) for people with Duffy null phenotype receiving treatment for multiple myeloma or triple negative breast cancer. The observational study is to collect dose modification and neutropenic fever information on patients who do not have the Duffy null phenotype and receive the same standard of care regimens to see if there are differences in dose modifications and neutropenic fever between the two groups. The survey studies seek to understand general health experiences and preferences and experiences specific to people with Duffy null phenotype.

Study Drugs Include:

* Daratumumab
* lenalidomide
* bortezomib
* dexamethasone
* carboplatin
* paclitaxel
* pembrolizumab
* cyclophosphamide
* doxorubicin

DETAILED DESCRIPTION:
This research study is a parallel arm, pragmatic, pilot study. As a pilot study it will be the first time investigators are examining using Duffy null specific dose modification guidelines for treatment dosing for participants with multiple myeloma or triple negative breast cancer receiving treatment of:

* Daratumumab, lenalidomide, bortezomib and dexamethasone for multiple myeloma
* Paclitaxel, carboplatin, doxorubicin, cyclophosphamide, and pembrolizumab for triple negative breast cancer The study will also be looking to understand health experiences of participants with and without the Duffy null phenotype through optional observational and survey studies.

The U.S. Food and Drug Administration (FDA) has approved daratumumab, lenalidomide, bortezomib and dexamethasone as a treatment option for some individuals with multiple myeloma. This study uses these drugs in ways typically used in clinical practice but not in ways approved by the FDA. Specifically, the FDA approval does not approve the use of this treatment for more than 4 cycles prior to stem cell transplantation or in those who are deferring or ineligible for transplantation, or with the specific drug dosing used in this study. These unapproved modifications, however, are supported by treatment guidelines from the National Comprehensive Cancer Network.

The U.S. Food and Drug Administration (FDA) has approved paclitaxel, carboplatin, doxorubicin, cyclophosphamide, and pembrolizumab for preoperative treatment of triple negative breast cancer. This study uses these drugs in ways typically used in clinical practice but not in ways approved by the FDA. Specifically, the FDA approval does not approve the use of this treatment in individuals who have 1-10% ER or PR positivity (called low-level positivity). This population, however, is often treated as having ER or PR negative disease, and this treatment decision is noted as acceptable by the National Comprehensive Cancer Network.

The research study procedures include screening for eligibility, clinical exams-medical history/physical exam, study treatment, and surveys.

The study treatment for the multiple myeloma group will be Bortezomib, Daratumumab, Lenalidomide, and Dexamethasone given over a 28 day cycle for 6 cycles.

The study treatment for the triple negative breast cancer group will receive treatment in two phases.

* The first phase will be Paclitaxel, carboplatin, and pembrolizumab over a 21 day cycle for 4 cycles.
* The second phase will be doxorubicin, cyclophosphamide, and pembrolizumab over a 21 day cycle for 4 cycles.

Participants who elect to take part in the optional observational studies will provide use of medical records for comparison of Duffy null and non-Duffy null populations. Participants who elect to take part in the optional short surveys will complete the short surveys.

It is expected that about 90 people will take part in this research study, 60 in the treatment study, and 30 in the observational study.

The Principal Investigator of this study and Dana-Farber Cancer Institute are the primary sponsors of this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of:

  * Cohort 1: MM, based on IMWG criteria12, and currently requires treatment
  * Cohort 2: Stage II or III TNBC, with definition per protocol Section 3.2.1 AND
* Plan for treatment, per their treating physician, or currently receiving their first cycle (see 3.3.3 for definition) of:

  * Cohort 1: Dara-RVd for MM
  * Cohort 2: A Keynote 522-based regimen of carboplatin, paclitaxel, and pembrolizumab given as the first phase of neoadjuvant treatment for TNBC.***

    * Participants are eligible even if the duration of carboplatin and paclitaxel goes beyond 4 cycles, or if the use of pembrolizumab, doxorubicin, and cyclophosphamide is not planned or is not certain, as long as neoadjuvant treatment starts with carboplatin-paclitaxel-pembrolizumab. This cohort will be referred to as "Keynote 522" for the remainder of the protocol.

AND

* Confirmed Duffy null phenotype

  * Previous testing is acceptable if performed by a CLIA-approved test

AND

* Age >=18 years old

Exclusion Criteria:

* Inability to understand and the willingness to sign a written informed consent document
* ANC<500 within 7 days of planned start of Cycle 1 Day 1.
* Participants who have started treatment at the time of enrollment cannot have started Cycle 2 of therapy
* Participants in Cohort 2 (TNBC) cannot have received any of the pembrolizumab, doxorubicin, and cyclophosphamide portion of therapy
* Participants receiving any other investigational agents for any indication
* Another known condition or medicine with known impacts on neutrophil counts or neutrophil function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Avoided or reduced systemic anticancer therapy (SACT) modifications per cycle | Avoided or reduced modifications determined by ANC (anticancer therapy) values in each treatment cycle. Coh 1 (Dara-RVD) is 6 cycles(cycle=28 dys)-ANC assessed days 1, 8, 15, & 22. Coh 2 has 8 cycles (cycle=21 dys)-ANC assessed days 1, 8, & 15
  An ANC-related avoided or reduced SACT change is defined as an instance of no change in SACT dosing (by avoiding a dose hold, dose level change, or drug discontinuation) OR an instance of reduction in the SACT dose modification (through earlier resumption of therapy with or without avoidance of a dose modification in a subsequent cycle) using this study's Duffy null-specific parameters for ANC dose modifications compared to the dose modification that would have occurred according to the parameters used in PERSEUS (Dara-RVD) or Keynote 522 trials. For the primary outcome measure, an ANC-related avoided or reduced SACT change is measured on a per-cycle basis as a binary outcome.
Overall cumulative incidence of neutropenic fever | Neutropenic fever is assessed from treatment initiation through the end of protocol-based treatment. It will be assessed at baseline and before treatment dosing during each cycle (Coh1 is 6 cycles (cycle=28 days); Coh 2 is 8 cycles (cycle=21 days)).
  Neutropenic fever is defined using modified CTCAE criteria. Grade 3 being defined as "ANC<500/uL with a single temperature of >38.3 C or a sustained temperature of >38 for more than one hour"; and Grade 4 defined as "Life-threatening consequences; urgent intervention indicated". The cumulative incidence will be calculated as the number of participants with at least one documented occurrence of neutropenic fever, over the total number of participants enrolled.

SECONDARY OUTCOMES:
Avoided or reduced systemic anticancer therapy (SACT) modifications per ANC check (i.e. per week) | Avoided or reduced modifications determined by ANC (anticancer therapy) values during each treatment cycle. Coh1 (Dara-RVD) is 6 cycles(cycle=28 dys)- ANC assessed on days 1, 8, 15, & 22. Coh 2 is 8 cycles (cycle=21 dys)- ANC assessed days 1, 8, & 15
  An ANC-related avoided or reduced SACT change is defined as an instance of no change in SACT dosing (by avoiding a dose hold, dose level change, or drug discontinuation) OR an instance of reduction in the SACT dose modification (through earlier resumption of therapy with or without avoidance of a dose modification in a subsequent cycle) using this study's Duffy null-specific parameters for ANC dose modifications compared to the dose modification that would have occurred according to the parameters used in PERSEUS (Dara-RVD) or Keynote 522 trials. For the secondary outcome measure, an ANC-related avoided or reduced SACT change is measured on a per-ANC check basis as a binary outcome.
Cumulative incidence of neutropenic fever within regimen | Neutropenic fever will be assessed from initiation of treatment through end of the last cycle of protocol-based treatment; cycle length and number varies by phase of therapy. It will be assessed at baseline and before therapy dosing during each cycle.
  Neutropenic fever is defined using modified CTCAE criteria. Grade 3 being defined as ""ANC<500/uL with a single temperature of >38.3 C or a sustained temperature of >38 for more than one hour""; and Grade 4 defined as ""Life-threatening consequences; urgent intervention indicated"". The cumulative incidence will be calculated as the number of participants with at least one documented occurrence of neutropenic fever, over the total number of participants enrolled in the regimen."
Relative dose intensity (RDI) | Dosing, for the calculation of RDI, will be assessed immediately at the time of protocol-specified treatment from the initiation of treatment through treatment completion, an average of 6 months. Cycle and treatment length vary by treatment phase.
  RDI will be calculated as the dose of the therapy administered divided by the dose as specified in the protocol. For multi-agent regimens, dose intensity will be calculated separately for each agent. Calculations will be done within patient.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hantel, MD, Principal Investigator — MD
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: andrew_hantel@dfci.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu